CLINICAL TRIAL: NCT04871048
Title: Examining tDCS Effect on Cannabis Use Disorder in Patients With Schizophrenia A Randomized Controlled Double-blind Exploratory Multicentric Study
Brief Title: Examining tDCS Effect on Cannabis Use Disorder in Patients With Schizophrenia
Acronym: CANNAPSYSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19PH229; 2020-A02976-33 (Other: ANSM)
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Cannabis-Induced Disorder
Keywords: dorsolateral prefrontal cortex; medial prefrontal cortex; schizophrenia; cannabis-induced disorder
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Stimulation will be performed using a Neurocan DC-Stimulator Plus with two 7×5 cm sponge electrodes soaked in a saline solution. Electrodes will be placed in accordance with the international 10-20 electrode placement system: the anode over F4 (right DLPFC), the cathode over Fp1 (MPFC). The stimulation level will be set at 2 mA for 20 minutes during stimulation sessions twice a day (separated by at least 3 hours) for 5 consecutive weekdays.
  The control group will receive the sham stimulation following the same regimen, using the sham procedure which has been developed by the manufacturer of the tDCS material, allowing sensations to be felt in the scalp which are the equivalent to those of the active stimulation. The same device will be used for both the sham and the active procedures.
Who Masked: Participant, Care Provider
Masking Description: * active tDCS stimulation. Patients will receive 10 sessions of tDCS over 5 consecutive days, at a frequency of 2 sessions per day spaced at least two hours apart, at an intensity of 2mA, for 20 minutes each.
  * tDCS placebo stimulation. Patients will receive 10 sessions of tDCS over 5 consecutive days, at a frequency of 2 sessions per day spaced at least two hours apart, following an identical procedure (tracking, then wearing the device for 20 minutes) but with actual stimulation provided during the first 40 seconds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS stimulation (Experimental): Transcranial direct current stimulation tDCS-Stimulation will be performed using a Neurocan DC-Stimulator Plus
  Interventions: Device: Transcranial direct current stimulation (tDCS) active
- sham tDCS stimulation (Sham Comparator): Transcranial direct current stimulation tDCS-The control group will receive the sham stimulation following the same regimen, using the sham procedure .
  Interventions: Device: Transcranial direct current stimulation (tDCS) non active

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) active — Stimulation will be performed using a Neurocan DC-Stimulator Plus with two 7×5 cm sponge electrodes soaked in a saline solution. Electrodes will be placed in accordance with the international 10-20 electrode placement system: the anode over F4 (right DLPFC), the cathode over Fp1 (MPFC). The stimulation level will be set at 2 mA for 20 minutes during stimulation sessions twice a day (separated by at least 3 hours) for 5 consecutive weekdays.
  Arms: active tDCS stimulation
Device: Transcranial direct current stimulation (tDCS) non active — The control group will receive the sham stimulation following the same regimen, using the sham procedure which has been developed by the manufacturer of the tDCS material, allowing sensations to be felt in the scalp which are the equivalent to those of the active stimulation. The same device will be used for both the sham and the active procedures.
  Arms: sham tDCS stimulation

SUMMARY:
Cannabis use disorder is a frequent comorbidity of schizophrenia, associated with increased symptoms and less adherence to therapy. Validated care has limited effectiveness in this population and development of new management strategies seems necessary. Transcranial direct current stimulation (tDCS) has shown beneficial effects in both schizophrenia, substance use disorder and, in a less extent, in nicotine addiction in schizophrenic subjects. It is interesting to test if that 10 sessions of anodal stimulation of the right dorsolateral prefrontal cortex (DLPFC) and cathodal stimulation of the medial prefrontal cortex (MPFC) (by increasing control and modulating reward system), will reduce, in 110 schizophrenic subjects, cannabis consumption, and secondly craving, addiction severity, schizophrenic symptoms and improve global functioning. It is possible that these clinical effects will be associated with changes in certain cognitive functions and cerebral connectivity.

DETAILED DESCRIPTION:
Stimulation will be performed using a Neurocan DC-Stimulator Plus with two 7×5 cm sponge electrodes soaked in a saline solution. Electrodes will be placed in accordance with the international 10-20 electrode placement system: the anode over F4 (right DLPFC), the cathode over Fp1 (MPFC). The stimulation level will be set at 2 mA for 20 minutes during stimulation sessions twice a day (separated by at least 3 hours) for 5 consecutive weekdays.

The control group will receive the sham stimulation following the same regimen, using the sham procedure which has been developed by the manufacturer of the tDCS material, allowing sensations to be felt in the scalp which are the equivalent to those of the active stimulation. The same device will be used for both the sham and the active procedures.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia diagnostic according to DSM (Diagnostic and Statistical Manual of mental disorder) 5 criteria, without change in psychotropic treatment since at least 4 weeks
* Moderate to severe cannabis use disorder according to DSM 5 criteria and active consumption during the last 7 days
* Subjects motivated to reduce or quit their cannabis consumption
* Patients with ambulatory compulsory care may be included

Exclusion Criteria:

* Other substance use disorder, excluding nicotine, according to DSM 5 criteria
* Other current psychiatric disorder according to DSM 5 criteria, excluding personality disorder
* Inpatient hospitalization
* History of head injury, neurological disorder with cerebral consequence or severe unstable somatic disorder
* Pregnancy or no contraception
* Contraindications for tDCS and/or MRI (implanted material, uncontrolled epilepsy, intracranial hypertension)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
cannabis use | 6 months
  Percentage change in cannabis use before and after tDCS treatment

SECONDARY OUTCOMES:
cannabis use | 3 months
  Percentage change in cannabis use before and after 3 months tDCS treatment
Change in craving scores | 3 months and 6 months
  Marijuana Craving Questionnaire score (minimum =12, maximum = 84). The higher the score, the greater the craving.
Hospitalizations | 6 months
  Number of hospitalization(s) during the 6 months after tDCS sessions
Study of structural cerebral connectivity | 3 months
  Cerebral MRI (only for a subgroup of patients) : Diffusion of water at the white matter level for the evaluation of structural brain connectivity in DTI mode (diffusion tensor) on
Study of structural and functional cerebral connectivity | 3 months
  Cerebral MRI (only for a subgroup of patients) : Functional connectivity index evaluated by resting state default mode network (MRI) for the evaluation of functional brain connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Aurelia GAY, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (8):
- France (8):
  - CH Le Vinatier Service universitaire d'addictologie de Lyon, Bron
  - Centre Hospitalier Universitaire Service d'Addictologie et Pathologies Duelles, Clermont-Ferrand
  - CHU de Clermont-Ferrand Service de Psychiatrie, Clermont-Ferrand
  - Service Hospitalo-Universitaire d'Addictologie CHU de Dijon, Dijon
  - CHU Pôle de Psychiatrie Neurologie et Rééducation, La Tronche
  - CH Saint-Cyr-au-Mont-d'Or service de psychiatrie, Saint-Cyr-au-Mont-d'Or
  - Centre Hospitalier Alpes Isère, Saint-Égrève
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No